CLINICAL TRIAL: NCT05954858
Title: Tissue Autograft to Bypass the Blood Brain Barrier (BBB) in Human Glioblastoma Multiforme (GBM)
Brief Title: Surgical Tissue Flap to Bypass the Blood Brain Barrier in Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0385
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioma, Malignant; Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme, Adult; High Grade Glioma; GBM; Brain Cancer
Keywords: tissue autograft; blood brain barrier; pedicled temporoparietal fascial; pericranial flap
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical tissue autograft: TPF flap/pericranial flap (Experimental): Use of a pedicled autologous piece of tissue called the temporoparietal fascial (TPF) flap or pericranial flap into the resection cavity of newly diagnosed glioblastoma multiforme (GBM) patients
  Interventions: Procedure: Tissue autograft of pedicled temporoparietal fascial (TPF) or pericranial flap to bypass the blood brain barrier (BBB)

INTERVENTIONS:
Procedure: Tissue autograft of pedicled temporoparietal fascial (TPF) or pericranial flap to bypass the blood brain barrier (BBB) — Surgical tissue autograft of pedicled temporoparietal fascial (TPF) or pericranial flap into the resection cavity of newly diagnosed glioblastoma multiforme (GBM) patients.
  Other Names: surgical tissue flap; tissue autograft

SUMMARY:
This single center, single arm, open-label, phase 2 study will assess the safety and efficacy of a pedicled temporoparietal fascial (TPF) or pericranial flap into the resection cavity of newly diagnosed glioblastoma multifome (GBM) patients.

The objective of the Phase 2 study is to demonstrate that this surgical technique is safe and effective in a human cohort of patients with resected newly diagnosed AA or GBM and may improve progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common primary central nervous system malignancy in adults, and accounts for over half of all malignant brain tumors. The prognosis for newly diagnosed GBM is extremely poor even with Stupp protocol consisting of surgery followed by temozolomide and radiotherapy. For newly diagnosed GBM the median overall survival (OS) is only 15 months, and the median progression-free survival (PFS) is a mere 5-6 months with only 53.9% of patients having 6 month PFS.

This Phase 2 study is an extension of our recently completely enrolled Phase I trial which showed the initial safety of a TPF into the resection cavity of newly diagnosed GBM. All 36 subjects included in this Phase 2 study will initially undergo standard surgical resection for newly diagnosed GBM. Following the resection, the surgical cavity will be lined with a long pedicled, autologous piece of tissue called a temporoparietal fascial flap or pericranium. The patient's dura, bone and scalp will be closed as is customary. The subject will be followed for side effects at 72 hours, 7 days, 30 days, 60 days, 120 days and 180 days. The primary outcome measure will be progression free survival (PFS) and secondary outcome measures will include overall survival (OS). Risk assessment will include seizure, stroke, infection, tumor progression, and death.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female 18 years of age or older.
2. Subject is undergoing planned resection of known or suspected GBM.
3. Subject has a Karnofsky Performance Status (KPS) 70% or greater.
4. Subject has a life expectancy of at least 6 months, in the opinion of the Investigator.
5. Based on the pre-operative evaluation by neurosurgeon, the subject is a candidate for ≥ 80% resection of enhancing region.
6. Subject must be able to undergo MRI evaluation.
7. Subject meets the following laboratory criteria:

   1. White blood count ≥ 3,000/μL
   2. Absolute neutrophil count ≥ 1,500/μL
   3. Platelets ≥ 100,000/μL
   4. Hemoglobin > 10.0 g/dL (transfusion and/or ESA allowed)
   5. Total bilirubin and alkaline phosphatase ≤ 2x institutional upper limit of normal (ULN)
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN
   7. Blood urea nitrogen (BUN) and creatinine < 1.5 x ULN
8. Females of reproductive potential must have a negative serum pregnancy test and be willing to use an acceptable method of birth control.
9. Males of reproductive potential must be willing to use an acceptable method of birth control to ensure effective contraception with partner.
10. Able to understand and willing to sign an institutional review board (IRB)- approved written informed consent document (legally authorized representative permitted).

Inclusion criteria considered during surgery:

1. Subject has a histologically confirmed (frozen section) diagnosis of WHO Grade IV glioblastoma multiforme (GBM).
2. TPFF and/or pericranial flap is technically feasible.

Exclusion Criteria:

1. Subject, if female, is pregnant or is breast feeding.
2. Subject has initiated chemotherapy or radiation treatment for diagnosis of or GBM.
3. Subject intends to participate in another clinical trial
4. Subject intends to undergo treatment with the Gliadel® wafer at the time of this surgery.
5. Subject has an active infection requiring treatment.
6. Subject has radiographic evidence of multi-focal disease or leptomeningeal dissemination.
7. Subject has a history of other malignancy, unless the patient has been disease- free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as localized prostate carcinoma or cervical carcinoma in situ after curative treatment
8. Subject has a known positive test for human immunodeficiency virus infection, or active hepatitis B or hepatitis C infection.
9. Subject has a history or evidence of any other clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  PFS is defined as time from surgery until first known disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS will be calculated as the time from treatment initiation (TPF implantation) to the time of death.

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Feinstein Institute for Medical Research/Lenox Hill Hospital
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No